CLINICAL TRIAL: NCT04011618
Title: Effect of Ellagic Acid Administration on the Components of Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion
Brief Title: Effect of Ellagic Ácid on the Components of Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Guadalajara (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Karina Griselda Pérez Rubio, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ellagic-SM
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Metabolic Syndrome
Keywords: ellagic acid; metabolic syndrome; insulin resistance; insulin secretion; insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Ellagic Acid

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: randomized double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 16 patients to receive 1 homologated placebo capsule (calcined magnesia 500 mg) every 12 hours along 12 weeks
  Interventions: Drug: Placebo oral capsule
- Ellagic acid (Experimental): 16 patients to receive 1 homologated intervention capsule (ellagic acid 500 mg) every 12 hours along 12 weeks
  Interventions: Drug: Ellagic Acid / Pomegranate Extract

INTERVENTIONS:
Drug: Ellagic Acid / Pomegranate Extract — Polyphenol, ellagitannin, it is found in a wide variety of fruits and nuts; in this particular case, pomegranate extract with 90% ellagic acid, 500 mg capsules. Homologated to the other intervention. Dosage twice a day orally every 12 hours during 12 weeks
  Other Names: benzoaric acid
  Arms: Ellagic acid
Drug: Placebo oral capsule — Calcined magnesia in 500mg capsules. Homologated to the other intervention. Dosage twice a day orally every 12 hours during 12 weeks
  Other Names: calcined magnesia
  Arms: Placebo

SUMMARY:
Metabolic syndrome (MetS) is a group of important cardiovascular risk factors: abdominal obesity, dyslipidemia, hyperglycemia, and high blood pressure. Treatment requires lifestyle changes and pharmacological therapy with different medications for each component. Ellagic acid (EA) is a polyphenol that has shown health benefits in multiple experimental studies. Patients consume EA without prescription; considering there aren't studies that demonstrate its effectiveness on MetS, it is important to evaluate the possible effects of AE on this pathology. METHODOLOGY: Current study is a double-blind, placebo-controlled clinical trial. The aim of this study is to evaluate the effect of AE on the components of metabolic syndrome, insulin sensitivity, and insulin secretion.

DETAILED DESCRIPTION:
INTRODUCTION: Ellagic acid (EA) is a polyphenol that has shown health benefits in multiple experimental studies; mainly as an antioxidant, but also in hepatic steatosis, endothelial damage, hypertension, diabetes mellitus, visceral fat accumulation, dyslipidemia, insulin resistance, atherosclerosis, etc. There aren't studies that demonstrate the effectiveness of EA on MetS; since patients consume it without any prescription, it is important to evaluate the effect of the administration of EA on the components of metabolic syndrome, insulin sensitivity, and insulin secretion. The current design is a randomized double-blind, placebo-controlled, clinical trial. METHODS: Male and female volunteers between 30 to 59 years of age, with a diagnosis of MetS according to the International Diabetes Federation criteria will be included, whether they accept participating and signing the informed consent. Patients with one or more of the following criteria will be excluded: History of liver, kidney, heart, or thyroid disease; diabetes mellitus or arterial hypertension, alcohol, drug abuse or tobacco use, systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg, fasting blood glucose ≥126 mg / dL, triglycerides ≥500 mg/dL, LDL cholesterol >190 mg/dL; suspected or confirmed pregnancy, lactation, menopausal period <1 year, hormonal contraceptive or replacement therapy, pharmacological, dietary or herbal therapy in the last 3 months before trial, allergy to any of the interventions. Patients included, may be withdrawn from the study if they meet any of the following conditions: Withdrawal of the informed consent, severe adverse reaction, loss of follow-up, treatment adherence <80%; intolerance to EA or placebo. OBJECTIVES: The main objective is to evaluate the effect of EA or placebo on metabolic syndrome components, insulin sensitivity, and insulin secretion. HEADQUARTERS: The study will be carried out in the facilities of the Institute of Experimental and Clinical Therapeutics (INTEC), of the University Center of Health Sciences, at the University of Guadalajara. Guadalajara, Jalisco, Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome diagnosis based on IDF criteria
* Acceptance and signing of Informed Consent

Exclusion Criteria:

* Prior diagnosis of kidney, liver, pancreas, heart or thyroid disease
* Diabetes mellitus or arterial hypertension
* Alcoholism, drug abuse or tobacco use
* Systolic blood pressure ≥140 mmHg
* Diastolic blood pressure ≥90 mmHg
* Fasting plasma glucose ≥126 mg/dL
* TG ≥500 mg/dL
* C-LDL > 190 mg/dL
* BMI: ≥35 kg/m2
* Pregnancy (suspected or confirmed) or lactation
* Menopausal period <1 year
* Hormonal contraceptive or replacement therapy
* Known allergy to any of the interventions
* Imposibility to shallow capsules
* Pharmacological, dietary or herbal therapy in the last 3 months before trial
* Weight variability above ±2.0 kg throughout the last 3 months before intervention

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
waist circunference | baseline to week 12 (end of intervention)
  Main criteria for metabolic syndrome diagnosis
blood pressure | baseline to week 12 (end of intervention)
  systolic blood pressure and diastolyc blood pressure by digital blood pressure monitor
fasting plasma glucose | baseline to week 12 (end of intervention)
  fasting plasma glucose by enzimatic-colorimetric automatized technique
Fasting plasma triglycerides | baseline to week 12 (end of intervention)
  fasting plasma triglycerides by enzimatic-colorimetric automatized technique
Fasting plasma HDL-c concentration | baseline to week 12 (end of intervention)
  fasting plasma high density lypoprotein-cholesterol by enzimatic-colorimetric automatized technique
Insulin sensitivity | baseline to week 12 (end of intervention)
  Estimated with Matsuda index. From an oral glucose tolerance test with glucose 75g intake, and each 30 minutes sampling to get insulin and glucose levels; minuted glucose and insulin results will be analized with Matsuda Index to get insulin sensitivity
Insulin secretion | baseline to week 12 (end of intervention)
  Stumvoll index will be used to calculate first-phase and area under curve (AUC) and ratio insulin AUC/glucose AUC for total insulin secretion

SECONDARY OUTCOMES:
body weight | baseline to week 12 (end of intervention)
  body weight measured by bioelectrical impedance scale
body mass index | baseline to week 12 (end of intervention)
  body mass index (BMI) calculated by Quetelet index
body fat mass | baseline to week 12 (end of intervention)
  body fat will be estimated by bioelectrical impedance analysis. Percentage.
Fasting plasma uric acid | baseline to week 12 (end of intervention)
  fasting plasma uric acid by enzimatic-colorimetric automatized technique
Fasting plasma insulin | baseline / week 12 (end of intervention)
  Fasting plasma insulin concentration by immunoassay
2 hours after oral-load glucose | baseline / week 12 (end of intervention)
  plasma glucose 2 hours after a 75 g oral glucose load
2 hours after oral-load insulin | baseline / week 12 (end of intervention)
  plasma insulin 2 hours after a 75 g oral glucose load
total cholesterol | baseline to week 12 (end of intervention)
  fasting plasma total cholesterol by enzimatic-colorimetric automatized technique
Fasting plasma LDL-c concentration | baseline to week 12 (end of intervention)
  fasting plasma low-density lipoprotein- cholesterol by enzimatic-colorimetric automatized technique
Fasting plasma VLDL concentration | baseline to week 12 (end of intervention)
  fasting plasma very low-density lipoprotein by enzimatic-colorimetric automatized technique
Concentration of plasma AST | baseline / week 12 (end of intervention)
  aminotransferases by enzimatic-colorimetric automatized technique
Concentration of plasma ALT | baseline / week 12 (end of intervention)
  aminotransferases by enzimatic-colorimetric automatized technique
Concentration of plasma creatinine | baseline / week 12 (end of intervention)
  creatinine by enzimatic-colorimetric automatized technique
Incidence of Adverse events related to placebo or ellagic acid | baseline to week 12 (continuous surveillance)
  Incidence of placebo or ellagic acid, emergent adverse events will be identified by clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: KARINA G PÉREZ-RUBIO, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- INSTITUTO DE TERAPÉUTICA EXPERIMENTAL Y CLÍNICA. Centro Universitario de Ciencias de la Salud, Guadalajara, Jalisco, Mexico